CLINICAL TRIAL: NCT05518773
Title: Mechanisms and Treatment of Exercise Intolerance and Persistent Fatigue in Spinal Muscular Atrophy
Status: Completed | Type: Observational
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Jacqueline Montes, Associate Professor of Rehabilitation and Regenerative Medicine, Rehab & Regenerative Med PT, Columbia University
Other Study IDs: AAAT5811
Record Dates: First submitted 2022-08-24; First posted 2022-08-29 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Spinal Muscular Atrophy
Keywords: spinal muscular atrophy; neuromuscular disease; risdiplam; nusinersen; aerobic capacity; oxygen uptake; fatigue; near infrared spectroscopy; muscle ultrasound; exercise tolerance; six minute walk test; mitochondria mitophagy; mitochondria; exercise; cycle ergometry; SMA
MeSH Terms: conditions — Muscular Atrophy, Spinal; Neuromuscular Diseases; Fatigue; Motor Activity | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Nusinersen treated: Children and adults who are currently treated with nusinersen for at least 6 months prior to enrollment.
  Interventions: Other: Observational
- Risdiplam treated: Children and adults who are currently treated with risdiplam for at least 6 months prior to enrollment.
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — Observational

SUMMARY:
This study will focus on the pathophysiological underpinnings of reduced exercise capacity and fatigue in ambulatory patients with spinal muscular atrophy (SMA). There has been laboratory evidence to suggest that the molecular mechanisms underlying mitochondrial biogenesis may be vulnerable to survival motor neuron (SMN) protein deficiency. This is an observational, single visit study including 34 ambulatory SMA patients treated with SMN repletion therapies (risdiplam or nusinersen) for at least 6 months at enrollment.

DETAILED DESCRIPTION:
SMN depletion affects muscle mitochondria and thus muscle function as a result. The relationship between these and their effect(s) on fatigue in the context of SMN repletion treatment has not been evaluated. If muscle function is vulnerable to SMN insufficiency, treatment strategies targeting muscle in addition to the central nervous system (motor neurons) may ameliorate fatigue and improve exercise capacity, thereby improving quality of life and bringing SMA treatments closer to a cure. This project explores such an idea by comparing the effects of the two different SMN repletion modalities in patients. This is an observational cross-sectional study involving ambulatory SMA children and adults treated for at least 6 months with SMN repletion therapy, either (1) systemically with risdiplam, or (2) intrathecally (central nervous system-only), with nusinersen.

ELIGIBILITY:
Inclusion Criteria:

* Genetic confirmation of SMA with laboratory documentation of homozygous deletion of survival motor neuron (SMN1) exon 7;
* At least 8 years of age at time of signing Informed Consent Form (or assent)
* Children or adults currently receiving treatment, for at least 6 months, with SMN repletion therapy, either with

  (1) risdiplam, or (2) nusinersen
* Able to walk independently at least 25 meters
* Able to tread a stationary cycle ergometer.

Exclusion Criteria:

* Unable to walk 25 meters independently.
* Use of investigational medications intended for the treatment of SMA within 30 days prior to study entry.
* The presence of any contraindication to exercise according the American College of Sports Medicine (ACSM) criteria.

Ages: 8 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study sample will include 34 ambulatory SMA patients, 17 currently treated with nusinersen, and 17 currently treated with risdiplam.
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2022-12-15 (Actual); Primary Completion 2025-11-14 (Actual); Study Completion 2025-11-14 (Actual)

PRIMARY OUTCOMES:
Peak oxygen uptake | Baseline
  Participants will undergo an exercise tolerance test performed by a clinical exercise physiologist using an electronically-braked recumbent cycle ergometer to determine peak oxygen uptake (VO2 max).

SECONDARY OUTCOMES:
NIRS derived index of muscle oxygen extraction | Baseline
  Near Infrared Spectroscopy (NIRS) is a simple, non-invasive method to measure oxygen in muscle and other tissues in vivo.
Distance walked during the Six Minute Walk Test (6MWT) | Baseline
  6MWT is an objective evaluation of functional exercise capacity, measures the maximum distance a person can walk in six minutes over a 25-meter linear course.
Leg muscle composition | Baseline
  To characterize leg muscle composition, quality and architecture using MRI and ultrasound in individuals with SMA treated with agents that restore SMN either systemically (risdiplam) or to central nervous system alone (nusinersen).

OTHER OUTCOMES:
Relationship of muscle quality and function | Baseline
  Muscle quality and architecture will be assessed using MRI and muscle ultrasound of the lower body, and the relationship to strength, function, and fitness will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Jacqueline Montes, PT, EdD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided